CLINICAL TRIAL: NCT02789917
Title: APixaban Versus PhenpRocoumon: Oral AntiCoagulation Plus Antiplatelet tHerapy in Patients With Acute Coronary Syndrome and Atrial Fibrillation
Brief Title: APixaban vs. PhenpRocoumon in Patients With ACS and AF: APPROACH-ACS-AF
Acronym: APPROACH
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: LMU Klinikum (Other)
Collaborators: Deutsches Zentrum für Herz-Kreislauf-Forschung (DZHK) (Other); Technical University of Munich (Other); Helmholtz Zentrum München (Industry); University of Göttingen (Other); University of München (Other); University Medicine Greifswald (Other)
Responsible Party: Principal Investigator, Reza Wakili, Professor Dr. med. Reza Wakili, LMU Klinikum
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GE IDE MucT003-16
Record Dates: First submitted 2016-05-24; First posted 2016-06-03 (Estimated); Last update posted 2020-08-14 (Actual); Status verified 2020-08

CONDITIONS: Acute Coronary Syndrome; Atrial Fibrillation; Coronary Artery Disease
Keywords: ACS; Triple-Therapy; AF; oral anticoagulation (OAC); non-vitamin-K oral anticoagulant (NOAC)
MeSH Terms: conditions — Acute Coronary Syndrome; Atrial Fibrillation; Coronary Artery Disease | interventions — Dual Anti-Platelet Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dual therapy (incl. NOAC) (Experimental): Apixaban plus Clopidogrel
  Interventions: Other: Dual Therapy
- Triple therapy (incl. VKA) (Active Comparator): Phrenprocoumon plus Clopidogrel plus ASA
  Interventions: Other: Triple Therapy

INTERVENTIONS:
Other: Dual Therapy — Combination of Apixaban 5mg/dl (or in reduced dosing of 2.5 mg/d depending on age, renal function and body weight) in combination with Clopidogrel 75 mg/d for 6 months.
  Arms: Dual therapy (incl. NOAC)
Other: Triple Therapy — HAS-BLED-Score <3:
  Combination of Phrenprocoumon (INR 2.0-2.5), Clopidogrel (75mg/d) and ASA (100 mg/d) for 6 months.
  HAS-BLED-Score ≥ 3:
  Combination of Phrenprocoumon (INR 2.0-2.5), Clopidogrel (75mg/d) and ASA (100 mg/d) for 1 month followed by Phrenprocoumon (INR 2.0-3.0) and Clopidogrel (75mg/d) for 5 months.
  Arms: Triple therapy (incl. VKA)

SUMMARY:
It is hypothesised that a dual therapy strategy by oral anticoagulation with the new Factor-Xa-inhibitor apixaban plus clopidogrel is superior to a triple therapy regimen with phenprocoumon plus acetylsalicylic acid (ASA) and clopidogrel with respect to avoiding bleeding events in patients with atrial fibrillation undergoing percutaneous coronary intervention in the setting of an acute coronary syndrome.

DETAILED DESCRIPTION:
Patients with atrial fibrillation (AF) presenting an acute coronary syndrome (ACS) and undergoing PCI require a triple therapy with a combination of oral anticoagulation (OAC) and dual anti-platelet therapy. Current guidelines recommend a regimen consisting of aspirin, clopidogrel and an oral anticoagulant. Although effective in preventing recurrent ischemia, triple therapy confers an elevated bleeding risk, which also has a major impact on the patients' prognosis and survival. Data from one randomized trial suggest that omitting aspirin in patients with indication for triple therapy may reduce the risk of bleeding without an increase of the rate of ischemic events. In addition, the recently introduced non-vitamin-K oral anticoagulants (NOACs) show less bleeding events as compared to vitamin-K antagonist in AF patients. In this trial it is postulated that a dual therapy consisting of the factor-Xa inhibitor apixaban and clopidogrel is associated with significant lower bleeding rates as compared to traditional triple therapy with aspirin, clopidogrel and a vitamin K antagonist (VKA). To test this hypothesis, patients with atrial fibrillation, who underwent PCI in the setting of an ACS will be randomized to either a dual therapy (apixaban+clopidogrel) or a triple therapy (aspirin+clopiodgrel+VKA). The patients will be followed-up for 6 months after randomization.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent
* Patients with an ACS after successful percutaneous coronary intervention
* Indication for oral anticoagulation due to non-valvular atrial fibrillation or atrial flutter (CHA2DS2VASc score ≥ 2)
* Males and Females, ages ≥ 18
* Women of childbearing potential (WOCBP) must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 24 hours prior to the start of study drug.
* Women must not be breastfeeding
* WOCBP must agree to follow instructions for method(s) of contraception for the duration of treatment with study drugs plus 30 days (duration of ovulatory cycle) post-treatment completion. However they must still undergo pregnancy testing.

Exclusion Criteria:

* Age < 18 years
* History of intracranial bleeding
* Active bleeding
* History of TIMI major bleeding according to TIMI and/or type ≥3b BARC criteria in the last 6 months
* History of peptic ulcer in the last 6 months
* Subjects with a history of a complicated or prolonged cardiogenic shock in the last two weeks prior to randomization. A complicated or prolonged cardiogenic shock is defined by a cardiogenic shock that required mechanical ventilation or the cardiovascular support with positive inotropic drugs (i.v. catecholamine) for ≥7 days
* Planned major surgery during the study course with planned discontinuation of antithrombotic therapy
* Expected life expectancy of less than a year and/or severe illness (e.g. malignancy)
* Mechanical valve replacement
* Valvular atrial fibrillation
* Severe renal insufficiency (creatinine clearance < 30ml/min)
* Severe liver insufficiency (Child-Pugh-class C) or elevated hepatic transaminases >2 times the upper limit of normal
* Patient's inability to fully comply with the study protocol
* Known or persistent abuse of medication, drugs or alcohol reliable by the investigator in individual cases
* Subjects with known contraindications to apixaban, phenprocoumon, clopidogrel or ASA treatment, which are hypersensitive to the drug substance or any component of the product
* Relevant hematologic deviations: platelet count < 50 G/L or platelet count > 600 G/L
* Current or planned pregnancy or nursing women, women 90 days after childbirth. Females of childbearing potential, who do not use and are not willing to use medically reliable methods of contraception for the entire study duration (such as oral, injectable, or implantable contraceptives, or intrauterine contraceptive devices) unless they are surgically sterilized / hysterectomized or there are any other criteria considered sufficiently

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 403 (Actual)
Dates: Start 2016-06; Primary Completion 2020-08 (Actual); Study Completion 2020-08 (Actual)

PRIMARY OUTCOMES:
The combined endpoint of moderate or major bleeding complications during the initial hospitalization and follow up (Bleeding Academic Research Consortium (BARC) type ≥ 2 bleeding) | up to 6 months after randomization

SECONDARY OUTCOMES:
Combined event of death, myocardial infarction, definite stent thrombosis, stroke/other systemic thromboembolism and all the individual components of the composite secondary endpoint | up to 6 months after randomization
Bleeding complications (Major bleeding: BARC > 3b bleeding) | up to 6 months after randomization

CONTACTS AND LOCATIONS:
Overall Officials: Reza Wakili, MD, Principal Investigator — Klinikum der Universität München (LMU); Steffen Massberg, Prof., Study Chair — Klinikum der Universität München (LMU)
Locations (16):
- Germany (16):
  - Munich University Hospital, Munich, Bavaria
  - Universitätsklinikum der RWTH Aachen, Aachen
  - Charité, Campus Benjamin Franklin, Berlin
  - Charité, Campus Virchow-Klinikum, Berlin
  - Klinikum Coburg, Coburg
  - Westdeutsches Herzzentrum am Universitätsklinikum, Essen
  - Universitätsmedizin Göttingen, Göttingen
  - Universitätsmedizin Greifswald, Greifswald
  - Universitätsklinikum Heidelberg, Heidelberg
  - UKHS Campus Kiel, Kiel
  - Klinikum Lüdenscheid, Lüdenscheid
  - Universitätsmedizin Mainz, Mainz
  - Universitätsklinikum Mannheim, Mannheim
  - Klinikum Augustinum, München
  - Städtisches Klinikum München-Neuperlach, München
  - Universitätsmedizin Rostock, Rostock

IPD SHARING:
Plan to Share IPD: Yes
Inclusion in central DZHK Database (German Centre for Cardiovascular Research)